CLINICAL TRIAL: NCT05557669
Title: Effect of Laparoscopic Cholecystectomy on Risk of Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brothers Hospitallers Hospital in Cracow (Other)
Collaborators: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Zofia Orzeszko, Principal Investigator, Brothers Hospitallers Hospital in Cracow
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1072.6120.25.2021
Record Dates: First submitted 2022-07-25; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Cholelithiasis; Metabolic Syndrome
MeSH Terms: conditions — Cholelithiasis; Metabolic Syndrome | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigation Group (Experimental): Patients undergoing laparoscopic cholecystectomy for cholelithiasis
  Interventions: Procedure: Laparoscopic cholecystectomy
- Control group (No Intervention): Patients with gallstone disease who are not planned for laparoscopic cholecystectomy in upcoming 3 months

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy is a procedure of removal of the gallbladder and a gold standard in treatment of gallstone disease.
  Arms: Investigation Group

SUMMARY:
Prospective cohort study. POPULATION: patients with gallstone disease qualified for laparoscopic cholecystectomy INTERVENTION: patients undergoing cholecystectomy for gallstones COMPARISON: gallstone disease without surgery in an observation period OUTCOME: metabolic syndrome symptoms evaluated in 3 months period The main inclusion criteria is cholelithiasis confirmed by ultrasound examination in patients between 18-75 years old. The main exclusion criteria are metabolic syndrome, diabetes, thyroid diseases, pancreatic diseases, serious abdominal surgeries in the past, pregnancy, and lactation. Participants who qualified for laparoscopic cholecystectomy in 3 months are included in the investigation group. Those not having cholecystectomy planned in the upcoming three months for any reason (no consent for surgery, long term) are included in the control group. The intervention is to assess all metabolic syndrome criteria (blood pressure, glucose tolerance, dyslipidemia, abdominal obesity) before and three months after surgery. The endpoint is to evaluate if the risk of metabolic syndrome after cholecystectomy is higher than in patients with gallstones.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is well known as a gold standard of treatment for gallstone disease. Gallbladder removal is one of the most common procedures in the United States, with more than 1.2 million cholecystectomies per year, and 92% of the procedures are performed laparoscopically. In 2011 Amigo et al. reported increased triglyceride levels in mice after cholecystectomy. According to Ruhl et al. (2013), cholecystectomy is associated with an increased risk of non-alcoholic fatty liver disease that is considered a liver manifestation of metabolic syndrome. In 2014, Shen et al. published a retrospective study enrolling 5672 participants that demonstrated an increased risk of metabolic syndrome after cholecystectomy compared with gallstone disease alone. Metabolic syndrome (MS) is a disease of civilization. It is a group of disorders containing impaired glucose intolerance, hypertension, abdominal obesity, and dyslipidemia. According to meta-analysis, individuals reaching the criteria of metabolic syndrome have a twice higher risk of myocardial infarction or stroke and a 1,5-times higher risk of death for any reason. The study aims to assess the risk of metabolic syndrome after laparoscopic cholecystectomy prospectively.

ELIGIBILITY:
Inclusion Criteria:

* cholelithiasis

Exclusion Criteria:

* metabolic syndrome
* obesity
* diabetes
* thyroid disease
* pancreatic disease
* serious abdominal surgeries in the past
* pregnancy, lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Risk of the metabolic syndrome in patients undergoing laparoscopic cholecystectomy | 3 months
  Evaluated with the rNCEP criteria for metabolic syndrome.
incidence of central obesity | 3 months
  waist circumference in cm: men more or equal 102 cm; women more or equal 88 cm
incidence of triglyceridemia | 3 months
  serum triglycerides level in mg/dl: more or equal 150 mg/dl
incidence of dyslipidemia | 3 months
  serum high-density lipo-protein (HDL) level in md/dl: men less than 40 mg/dl; women less than 50 mg/dl
incidence of systemic hypertension | 3 months
  blood preassure in mm Hg: more or equal 130 mm Hg/more or equal 85 mm Hg
incidence of glucose intolerance | 3 months
  fasting serum glucose in mg/dl: more or equal 100 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Mirosław Szura, prof., Study Chair — Jagiellonian University
Locations (1):
- Brothers Hospitallers Hospital in Cracow, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrera F, Azocar L, Molina H, Schalper KA, Ocares M, Liberona J, Villarroel L, Pimentel F, Perez-Ayuso RM, Nervi F, Groen AK, Miquel JF. Effect of cholecystectomy on bile acid synthesis and circulating levels of fibroblast growth factor 19. Ann Hepatol. 2015 Sep-Oct;14(5):710-21. PMID 26256900
- [Background] Latenstein CSS, Alferink LJM, Darwish Murad S, Drenth JPH, van Laarhoven CJHM, de Reuver PR. The Association Between Cholecystectomy, Metabolic Syndrome, and Nonalcoholic Fatty Liver Disease: A Population-Based Study. Clin Transl Gastroenterol. 2020 Apr;11(4):e00170. doi: 10.14309/ctg.0000000000000170. PMID 32352682
- [Background] Chen Y, Wu S, Tian Y. Cholecystectomy as a risk factor of metabolic syndrome: from epidemiologic clues to biochemical mechanisms. Lab Invest. 2018 Jan;98(1):7-14. doi: 10.1038/labinvest.2017.95. Epub 2017 Sep 11. PMID 28892095
- [Background] Di Ciaula A, Garruti G, Wang DQ, Portincasa P. Cholecystectomy and risk of metabolic syndrome. Eur J Intern Med. 2018 Jul;53:3-11. doi: 10.1016/j.ejim.2018.04.019. Epub 2018 Apr 26. PMID 29706426
- [Background] Garruti G, Wang DQ, Di Ciaula A, Portincasa P. Cholecystectomy: a way forward and back to metabolic syndrome? Lab Invest. 2018 Jan;98(1):4-6. doi: 10.1038/labinvest.2017.129. PMID 29297503
- [Background] Qi L, Tian Y, Chen Y. Gall bladder: The metabolic orchestrator. Diabetes Metab Res Rev. 2019 Jul;35(5):e3140. doi: 10.1002/dmrr.3140. Epub 2019 Feb 27. PMID 30770629
- [Background] Tsai MS, Lin CL, Hsu YC, Lee HM, Kao CH. Long-term risk of pancreatitis and diabetes after cholecystectomy in patients with cholelithiasis but no pancreatitis history: a 13-year follow-up study. Eur J Intern Med. 2015 Sep;26(7):540-4. doi: 10.1016/j.ejim.2015.06.013. Epub 2015 Jul 2. PMID 26143191
- [Background] Yue W, Sun X, Du T. Cholecystectomy versus central obesity or insulin resistance in relation to the risk of nonalcoholic fatty liver disease: the third US National Health and Nutrition Examination Survey. BMC Endocr Disord. 2019 Sep 2;19(1):95. doi: 10.1186/s12902-019-0423-y. PMID 31477078